CLINICAL TRIAL: NCT07330739
Title: Kinesiophobia in Women With Stress Urinary Incontinence
Status: Active, not recruiting | Type: Observational
Sponsor: Esra BAYRAMOĞLU DEMİRDÖĞEN (Other)
Responsible Party: Sponsor-Investigator, Esra BAYRAMOĞLU DEMİRDÖĞEN, LECTURER DOCTOR, Ahi Evran University Education and Research Hospital
Organization: Ahi Evran University Education and Research Hospital (Other)
Other Study IDs: KAEU-EBAYRAMOGLUD-005
Record Dates: First submitted 2025-12-21; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Kinesiophobia
MeSH Terms: conditions — Kinesiophobia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stress Urinary Incontinence
  Interventions: Other: Survey
- Control
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — survey

SUMMARY:
All women included in the study will be administered the Causes of Kinesiophobia Scale (KCS), the International Physical Activity Questionnaire (Short), the International Incontinence Consultation Questionnaire-Short Form (ICIQ-SF), and the Pittsburgh Sleep Quality Questionnaire (PSQI). Subsequent analysis will determine the causes of kinesiophobia in women with urinary incontinence.

DETAILED DESCRIPTION:
All women included in the study will be administered the Causes of Kinesiophobia Scale (KCS), the International Physical Activity Questionnaire (Short), the International Incontinence Consultation Questionnaire-Short Form (ICIQ-SF), and the Pittsburgh Sleep Quality Questionnaire (PSQI). Subsequent analysis will determine the causes of kinesiophobia in women with urinary incontinence. The results will then be compared with those of healthy women.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18-65 years old
2. Having stress urinary incontinence
3. Voluntary participation in the study

Exclusion Criteria:

1. Unwillingness to continue working
2. Presence of neurological or orthopedic disease
3. Learning disability or other cognitive impairments.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women with stress urinary incontinence
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | day 1
  Kinesiophobia, or fear of movement, in patients will be assessed using the Causes of Kinesiophobia Scale. This scale consists of 20 questions and evaluates the fear of movement in two subcategories: biological and psychological causes.

CONTACTS AND LOCATIONS:
Overall Officials: ESRA bayramoğlu demirdöğen, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kirşehir Ahi Evran University Physical Therapy and Rehabilitation Hospital, Kırşehir, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No